CLINICAL TRIAL: NCT00542867
Title: Pan-European Survey on the Under Treatment of Hypercholesterolemia
Acronym: CEPHEUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: SRP-CB-CRE-2006/01
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Third Joint European Task Force guidelines; Survey
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The survey try to establish the proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the Third Joint European Task Force guidelines, overall and by country.·

ELIGIBILITY:
Inclusion Criteria:

* Patients had to be on a lipid-lowering drug treatment for at least 3 months, with no dose change for a minimum of 6 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6500 (Actual)
Dates: Start 2006-01; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The number and percentage of patients achieving the LDL-C goals, according to the Third Joint European Task Force guidelines, overall and by country.

CONTACTS AND LOCATIONS:
Overall Officials: M. Hermans, Principal Investigator — UCL

REFERENCES:
- [Derived] Hermans MP, Castro Cabezas M, Strandberg T, Ferrieres J, Feely J, Elisaf M, Michel G, Sansoy V. Centralized Pan-European survey on the under-treatment of hypercholesterolaemia (CEPHEUS): overall findings from eight countries. Curr Med Res Opin. 2010 Feb;26(2):445-54. doi: 10.1185/03007990903500565. PMID 20001658